CLINICAL TRIAL: NCT06916819
Title: Food Challenge at Home or in Medical Practice - a Multi-center Randomized Control Trial - FoodCHOMP Study
Brief Title: Food Challenge at Home or in Medical Practice - the FoodCHOMP Study
Acronym: CHOMP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Austin Health (Other Government)
Collaborators: Royal Melbourne Hospital, Australia (Unknown)
Responsible Party: Principal Investigator, Jack Godsell, Dr Jack Godsell, Clinical Immunologist and Allergist, Principal Investigator, Austin Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 111750/Austin-2024
Record Dates: First submitted 2025-03-26; First posted 2025-04-08 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Food Allergies
Keywords: Food allergy; Food allergy label; Food Challenge
MeSH Terms: conditions — Food Hypersensitivity

STUDY DESIGN:
Intervention Model Description: This study uses a parallel assignment model. Participants who meet eligibility criteria are randomly assigned in a 1:1 ratio to one of two arms: a home-based food challenge group (intervention) or a standard in-clinic food challenge group (control). Each participant undergoes only one of the two interventions, and there is no crossover between arms. Randomisation is stratified by site and gender and conducted via REDCap using a permuted block design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- In-Clinic Food Challenge (Control Arm) (Other): Participants randomised to the control arm will undergo a standard in-clinic oral food challenge conducted under direct medical supervision. The protocol used is derived from the PRACTALL consensus and ASCIA position statements and involves administration of increasing doses of the implicated food at 20-30 minute intervals over a 2-3 hour period. Observation continues for 1-2 hours post final dose. The challenge is performed in a hospital outpatient clinic equipped for anaphylaxis management. The food challenged is selected by the participant from their eligible food allergy labels.
  Interventions: Diagnostic Test: In-Clinic Food Challenge
- Home-Based Food Challenge (Intervention Arm) (Experimental): Participants randomised to the intervention arm will undertake a structured home-based oral food challenge over five consecutive days. This begins with an initial supervised dose administered in clinic under medical observation (60-minute monitoring period). Participants will then self-administer increasing doses of the implicated food at home each subsequent day using a standardised protocol adapted from PRACTALL and ASCIA guidelines. Dose intervals are 24 hours to reduce risk of cumulative reactions. Participants are provided with written instructions, emergency action plans, and have daily phone follow-up with allergy nursing staff during the challenge. The challenge food is selected by the participant from their eligible food allergy labels.
  Interventions: Diagnostic Test: Home-Based Food Challenge

INTERVENTIONS:
Diagnostic Test: Home-Based Food Challenge — Participants randomised to the intervention arm will undertake a structured home-based oral food challenge over five consecutive days. This begins with an initial supervised dose administered in clinic under medical observation (60-minute monitoring period). Participants will then self-administer increasing doses of the implicated food at home each subsequent day using a standardised protocol adapted from PRACTALL and ASCIA guidelines. Dose intervals are 24 hours to reduce risk of cumulative reactions. Participants are provided with written instructions, emergency action plans, and have daily phone follow-up with allergy nursing staff during the challenge. The challenge food is selected by the participant from their eligible food allergy labels.
  Arms: Home-Based Food Challenge (Intervention Arm)
Diagnostic Test: In-Clinic Food Challenge — Standard of care - Participants randomised to the control arm will undergo a standard in-clinic oral food challenge conducted under direct medical supervision. The protocol used is derived from the PRACTALL consensus and ASCIA position statements and involves administration of increasing doses of the implicated food at 20-30 minute intervals over a 2-3 hour period. Observation continues for 1-2 hours post final dose. The challenge is performed in a hospital outpatient clinic equipped for anaphylaxis management. The food challenged is selected by the participant from their eligible food allergy labels.
  Arms: In-Clinic Food Challenge (Control Arm)

SUMMARY:
This is a pilot, multi-centre, randomised clinical trial evaluating the safety and feasibility of a home-based oral food challenge in adults with low-risk food allergy labels. Eligible participants are aged 18 years or older and have a self-reported food allergy with negative skin prick testing to the implicated food. Participants will be randomised to either a home-based or standard in-clinic food challenge. The primary aim is to determine the safety of home challenges, measured by the rate of immune-mediated adverse events. Secondary aims include feasibility of recruitment and delivery, protocol adherence, quality of life, and food reintroduction outcomes.

DETAILED DESCRIPTION:
Food allergies are highly prevalent and contribute to significant patient anxiety and healthcare utilisation. Many individuals carry food allergy labels without confirmation through diagnostic food challenge, resulting in unnecessary food avoidance. In-clinic food challenges are the current standard for confirming tolerance but are resource-intensive and often delayed. This study evaluates whether selected low-risk adults can safely complete a structured oral food challenge at home.

This is a pilot, multi-centre, randomised controlled trial conducted at two tertiary allergy centres in Victoria, Australia (Austin Health and Royal Melbourne Hospital). Adults referred with a reported food allergy will undergo clinical assessment and skin prick testing. Those with negative skin testing (<3mm wheal) to the implicated food and meeting other eligibility criteria will be randomised 1:1 to either:

* Intervention: Home-based oral food challenge over five days, beginning with a single supervised dose in-clinic and followed by four incremental doses at home with daily clinical follow-up.
* Control: Standard in-clinic oral food challenge using a protocol derived from PRACTALL and ASCIA guidelines.

The primary outcome is the proportion of participants experiencing an immune-mediated adverse event during food challenge. Secondary outcomes include feasibility metrics (eligibility, recruitment, delivery), non-immune mediated adverse events, protocol adherence, quality of life (measured by FAQLQ-12), time to challenge, and real-world food reintroduction.

The study will enrol 120 participants (60 per arm). Outcomes will inform the design of a future non-inferiority trial and may support integration of home challenges into routine practice for selected patients.

ELIGIBILITY:
Inclusion Criteria:

1. Negative (<3mm) fresh or extract skin testing to the food implicated within their allergy label
2. Aged greater than 18 years

Exclusion Criteria:

* Evidence of prior sensitisation to challenge food 0 Defined as previously positive skin testing or allergen specific IgEs if available
* Pregnancy
* Patients with poorly controlled asthma - defined as an ACQ5 scores >1 at the time of enrolment
* Patients with a history of food reactions that is not-consistent with an IgE mediated process; i.e. exclusively gastrointestinal symptoms, FPIES
* Patients with a clear history of food-dependent exercise induced anaphylaxis
* Patients on a concurrent medication which may influence the outcome of the challenge;
* Antihistamine therapy; Patients receiving more than stress dose steroids (i.e. > 50mg QID hydrocortisone [or steroid equivalent]); Omalizumab
* Any other illness that, in the investigator's judgement, will substantially increase the risk associated with subject's participation in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2025-04-16 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants experiencing immune-mediated adverse events during food challenge | During the food challenge period (Days 1-5 post-randomisation)
  Immune-mediated adverse events are defined as clinical symptoms consistent with IgE-mediated food allergy occurring during the food challenge, including but not limited to: urticaria, angioedema, vomiting, diarrhoea, or respiratory compromise (e.g., wheezing, cough, stridor). Events will be recorded according to a standardised adverse event form. For home challenges, participants will self-report symptoms daily and receive follow-up via nursing staff. In-clinic events will be recorded by supervising clinicians.

SECONDARY OUTCOMES:
Proportion of screened patients who are eligible for randomisation (Eligibility-to-screened ratio) | Baseline visit
  Feasibility metric defined as the proportion of patients referred to outpatient allergy clinic who meet the trial eligibility criteria (including negative skin prick testing to the implicated food and absence of exclusion criteria).
Proportion of eligible patients who consent to participate (Recruitment-to-eligibility ratio) | At consent discussion (baseline visit)
  Feasibility of recruitment measured as the proportion of eligible patients who provide written informed consent to participate in the trial.
Proportion of randomised participants who receive the allocated intervention (Intervention-to-recruitment ratio) | Day 1 to Day 5 (intervention delivery period)
  Defined as the proportion of randomised participants who complete their allocated food challenge (home or in-clinic) in accordance with protocol.
Proportion of participants experiencing non-immune mediated adverse events | Day 1 to Day 5 (challenge period)
  Non-immune mediated events include those not consistent with IgE-mediated allergy and not meeting serious adverse event criteria. Examples: taste aversion, food refusal, procedural anxiety. Events will be recorded via self-report or in-clinic observation.
Proportion of participants with severe adverse reactions (anaphylaxis or death) | Day 1 to Day 5 (challenge period)
  Serious adverse events are defined per ICH-GCP and include anaphylaxis (as per ASCIA criteria) or death.
Difference in proportion of participants tolerant to challenge food | At completion of challenge (Day 5)
  Defined as the proportion of participants in each arm who successfully consume the full challenge dose without meeting stopping criteria or experiencing adverse events. Tolerance is determined according to protocol-defined thresholds.
Change in Food Allergy Quality of Life (FAQLQ-12) score from baseline | Baseline and 6 months post-randomisation
  Measured using the FAQLQ-12, a validated 12-item quality of life tool for adults with food allergy. Change in score will be assessed as a continuous variable.
Proportion of participants consuming the challenge food post-trial | At 6-month follow-up
  Defined as the proportion of participants who report active inclusion of the challenge food in their diet at least once per week following a successful challenge.
Time from clinic referral to challenge completion | From the date of referral for food challenge to date of challenge completion or withdrawal from the study assessed up to 60 months.
  Measured in days to assess whether home-based challenge reduces diagnostic delay compared to in-clinic challenge.
  Data collected through clinic administrative records.

CONTACTS AND LOCATIONS:
Locations (2):
- Australia (2):
  - Austin Health, Melbourne, Victoria
  - Royal Melbourne Hospital, Melbourne, Victoria

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD with other researchers

REFERENCES:
- [Derived] Godsell J, Vogrin S, Chan S, Henri M, Ng I, Andrews E, Spriggs K, Perrett KP, Trubiano J. FoodCHOMP (Food Challenge-at HOme or in Medical Practice): a pilot multicentre randomised controlled trial evaluating home versus clinic-based food allergy challenges in low-risk adults-study protocol. BMJ Open. 2026 Feb 6;16(2):e114483. doi: 10.1136/bmjopen-2025-114483. PMID 41651530